CLINICAL TRIAL: NCT01409291
Title: Impact of a Financial Success Education Program on Perceived Financial Well-being, Hopefulness, Financial Competency, Financial Goal Achievement, Quality of Life, and Quantitative Health Outcomes in Women and Children: A Pilot Study
Brief Title: Impact of a Financial Success Education Program in Women and Children
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-16171
Record Dates: First submitted 2011-07-29; First posted 2011-08-04 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Stress
Keywords: low socioeconomic status; stress; women; children; cortisol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many Americans are living paycheck to paycheck. This may lead to financial stress and an increase in overall stress. People under stress are more likely to smoke, consume alcohol, eat a poor diet, and experience depression or anxiety. Experiencing financial stress may also increase the risk for heart disease. The purpose of this research study is to test whether participating in the Financial Success Program improves health outcomes, in both the women participating and their children.

ELIGIBILITY:
Inclusion Criteria:

* Women 19 years or older enrolled in the Financial Success Program in fall 2011 and winter 2012 and/or a their child(ren) ages 3-18 years attending the daycare with their mother
* Women must be employed to be enrolled in the Financial Success Program
* Able and willing to provide informed consent

Exclusion Criteria:

* Women less than 19 years of age
* Women working a night time shift (due to variability in diurnal cortisol secretion)
* Known pregnancy or planned pregnancy (due to variability in blood pressure, glucose, weight, and lipids)
* Women are excluded from the Financial Success Program if they are living in a domestic violence situation or abusing alcohol or illicit drugs

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women enrolled in the Financial Success Program and their children
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Packard, PharmD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Result] Packard KA, Kalkowski J, White N, Ryan-Haddad A, Black L, Flecky K, Furze J, Rusch L, Qi Y. Chapter 5: Impact of a financial education program in single, low-income women and their children. In: Public Health: Improving Health via Inter-Professional Collaborations Ed: Rosemary M. Caron and Joav Merrick. 2014.
- [Result] White N, Packard KA, Kalkowski J, Ryan-Haddad A, Flecky K, Furze J, Rusch L, Black L. Chapter 6: A novel financial education program in single women of low-income and their children In: Public Health: Improving Health via Inter-Professional Collaborations Ed: Rosemary M. Caron and Joav Merrick. 2014.

RESULTS

PARTICIPANT FLOW:
Groups:
- Mothers: All participants of the Financial Success Program were approached for the study. This was a single arm descriptive study.
- Children: Children between ages 3 and 18 years whose mothers were participating in the Financial Success Program.
Period: Overall Study
Arm/Group | Mothers | Children
Started | 36 | 28
Completed | 29 | 19
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mothers | Children | Total
Number analyzed (Participants) | 36 | 28 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (6.1) | 7.9 (3.5) | 23.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 16 | 52
  Male | 0 | 12 | 12
Region of Enrollment [Number; unit: participants]
  United States | 36 | 28 | 64

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Exercise Per Week
Description: Mean minutes of exercise per week
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Mothers | Children
Number analyzed (Participants) | 36 | 28
minutes
  Pre-intervention | 120.0 (237.0) | 404.5 (319.6)
  1-year | 184.2 (404.2) | 350.3 (246.8)

2. Secondary Outcome: Fast Food Meals Per Week
Description: Mean number of fast food meals per week
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: meals per week
Arm/Group | Mothers | Children
Number analyzed (Participants) | 36 | 28
meals per week
  Pre-intervention | 2.4 (1.7) | 1.9 (1.4)
  1-year | 1.5 (1.1) | 1.4 (1.3)

ADVERSE EVENTS:
Arm/Group | Mothers | Children
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/26
Other Adverse Events (participants affected / at risk) | 0/38 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes